CLINICAL TRIAL: NCT02223403
Title: Single Dose of Nitrate-rich Beetroot Juice Does Not Improve Steady State Oxygen Consumption or Six-minute Walk Distance in Patients With Systolic Heart Failure.
Brief Title: Effect of Nitrate-rich Beetroot Juice on Exercise Performance in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth M Leclerc, MD, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 383967-4
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Systolic Heart Failure
Keywords: Nitrate-rich beetroot juice; heart failure; exercise performance; oxygen consumption
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- submaximal steady state exercise (Experimental): 90 minutes after respective beetroot juice ingestion, subjects walked on treadmill at a pre-determined steady state workload for a total of 15 minutes with oxygen consumption recorded for the last 10 minutes
  Interventions: Dietary Supplement: nitrate-rich beetroot juice; Dietary Supplement: nitrate-deplete beetroot juice
- six minute walk test (Experimental): subjects performed six-minute walk at self-determined pace 30 minutes after treadmill exercise was performed
  Interventions: Dietary Supplement: nitrate-rich beetroot juice; Dietary Supplement: nitrate-deplete beetroot juice

INTERVENTIONS:
Dietary Supplement: nitrate-rich beetroot juice — 3 ounces of nitrate-rich beetroot juice ingested orally once 90 minutes before exercise interventions of steady state treadmill exercise followed 30 minutes later by six minute walk
  Other Names: Beet It Sport Stamina Shot
Dietary Supplement: nitrate-deplete beetroot juice — 3 ounces of nitrate-deplete beetroot juice ingested orally once 90 minutes before exercise interventions of steady state treadmill exercise followed 30 minutes later by six minute walk
  Other Names: Beet It Sport Stamina Shot

SUMMARY:
Nitrate-rich beetroot juice supplementation has demonstrated reduced oxygen consumption and submaximal exercise performance in healthy adults. Investigation for similar effects in patients with heart failure has not previously been conducted.

This was a randomized, double-blind, placebo controlled trial. Following ingestion of the active agent or placebo, subjects with systolic heart failure underwent submaximal steady state exercise with gas exchange analysis followed thirty minutes later by a six minute walk test. Second testing sessions were performed ten days.

There were no significant differences in the treatment and placebo arms in average oxygen consumption or six minute walk distance.

In conclusion, in patients with heart failure who have ingested a single dose of nitrate-rich beetroot juice concentrate, there is no significant difference with regard to oxygen consumption during submaximal steady state exercise or six minute walk testing distance.

Further study is warranted to determine the true efficacy of nitrate consumption in this population with adjustments in acute or chronic dosing, exercise duration, or intensity.

ELIGIBILITY:
Inclusion Criteria:

* Local institutional beneficiaries between the ages of 18 and 80
* Documentation of left ventricular systolic dysfunction with ejection fraction < 40% by any modality within the past six months
* Documentation of New York Heart Association class II or III status.

Exclusion Criteria:

* > 80 years of age
* Unable to adequately or safely perform treadmill exercise
* Pulmonary disease deemed significant enough to be a limitation to exercise
* Greater than moderate stenotic or regurgitant valvular heart disease
* Presence of atrial fibrillation or other uncontrolled arrhythmias
* Uncompensated heart failure
* Continuously paced rhythms
* Pregnant females
* Chronic nitroglycerine use (oral isosorbide di or mono-nitrate, or topical nitroglycerine)
* Phosphodiesterase inhibitor (sildenafil or tadalafil) use within a week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
steady state exercise oxygen consumption | 10 minutes
  Subjects performed steady state treadmill walking at a pre-determine submaximal workload. Oxygen consumption was measured for the last 10 minutes.
six minute walk distance | six minutes
  subjects walked at their chosen pace for six minutes on a pre-determined course. Total distance was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Leclerc, MD, Principal Investigator — Brooke Army Medical Center